CLINICAL TRIAL: NCT04839250
Title: Study on The Difference Between Three-Dimensional Heads-Up Surgery System and Traditional Surgery Methods in Cataract Surgery
Brief Title: Difference Between Three-Dimensional Heads-Up Surgery System and Traditional Surgery Methods in Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Yune Zhao, Vice president of Eye Hospital of Wenzhou Medical University, Wenzhou Medical University, Wenzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3D system-CPJ
Record Dates: First submitted 2021-04-04; First posted 2021-04-09 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Cataract
Keywords: three-dimensional surgery; microsurgery; phacoemulsification
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cataract surgery performed by heads-up method (Experimental): 3D heads-up surgery was performed under the NGENUITY® 3D visualization system
  Interventions: Procedure: heads-up method
- Traditional surgery (No Intervention): Traditional surgery was performed under a surgical microscope.

INTERVENTIONS:
Procedure: heads-up method — 3D surgical video system, which includes Alcon NGENUITY 3D visualization system (Alcon, Fort Worth, TX) and Leica M822 and M844 microscopes (Leica Microsystems, Wetzlar, Germany),can be used to perform head-up phacoemulsification combined with intraocular lens implantation surgery.
  Arms: cataract surgery performed by heads-up method

SUMMARY:
To evaluate the differences between three-Dimensional heads-Up surgery system and traditional surgery methods of cataract surgery

DETAILED DESCRIPTION:
To evaluate the differences between three-Dimensional heads-Up surgery system and traditional surgery methods of cataract surgery.Prospective research.One eligible eye from patients having cataract surgery performed using the 3-D head-up technique were included in the study as an experimental group,in the meanwhile eyes performed cataract surgery by traditional microsurgery included as a control group.All eyes in the study are operated by the same doctor. Corneal incision form,corneal endothelial cell density and best corrected visual acuity are included to evaluate the results of cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnose age-related cataract;
2. Plan to perform phacoemulsification of cataract with intraocular lens implantation;
3. Willing to cooperate with the re-examination of 1 day, 1 week, and 1 month after surgery;
4. Able to understand and independently fill in the informed consent form and postoperative follow-up plan.

Exclusion Criteria:

1. Cataract caused by other reasons;
2. Fundus diseases such as severe diabetic retinopathy, high myopic retinopathy or macular degeneration;
3. Corneal diseases, corneal endothelial cells <1800/mm2;
4. Small palpebral fissure;
5. Those with a history of glaucoma, uveitis, eye trauma or eye surgery;
6. Those who cannot cooperate with the inspection and have not completed the one-month follow-up

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
change of corneal incision from 1day after surgery to 1 months | up to 1day,1week,1 month
  the shape and length of the corneal incision ，if descemet's layer detachment happens
corneal endothelial cell density | up to 1 month
  the number of corneal endothelial cells per unit area

SECONDARY OUTCOMES:
best corrected visual acuity | up to 1 month
  best corrected visual acuity
change from baseline central corneal thickness at 1 months | up to 1 day,1 week,1 month
  thickness in micrometer
change from baseline corneal incision thickness at 1 months | up to 1 day,1 week,1 month
  Thickness of corneal incision

CONTACTS AND LOCATIONS:
Locations (1):
- Eye Hospital of Wenzhou Medical College, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhu Z, Chang P, Huang F, Shen S, Zhao X, Ji X, Zhao YE. Comparison of Three-Dimensional Surgical System Versus Binocular Microscope for Clear Corneal Incision in Cataract Surgery. Ophthalmol Ther. 2022 Aug;11(4):1589-1600. doi: 10.1007/s40123-022-00537-4. Epub 2022 Jun 24. PMID 35749016